CLINICAL TRIAL: NCT05997394
Title: The Effect of Prayer on Dyspnea Severity, Anxiety and Spiritual Well-Being in Individuals With COPD
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Gülden Kaygusuz, Graduate Student, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCU-SBF-GK-01
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: COPD
Keywords: DYSPNEA; SPIRITUAL GOODNESS; ANXIETY
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: It is a semi-experimental type of study. It consists of two groups: experiment and control.
Who Masked: Participant, Investigator
Masking Description: The experimental and control groups will be determined by randomization method by a person other than the researcher. Participants will not know which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in this group will be given a prayer concert for a month. At the end of one month, the severity of dyspnea, anxiety and spiritual well-being levels experienced by the participants will be re-checked.
  Interventions: Other: A prayer concert will be held for the participants.
- Control Group (No Intervention): There will be no prayer audience for participants in this group.

INTERVENTIONS:
Other: A prayer concert will be held for the participants. — Participants who are in the experimental group will be given a prayer audience.
  Arms: Experimental Group

SUMMARY:
This study will be conducted in order to examine the effect of prayer to individuals with COPD on the severity of dyspnea, anxiety and spiritual well-being experienced by patients.

DETAILED DESCRIPTION:
This study will be conducted on people with COPD. People with COPD disease will be divided into two groups. The experimental group will be given a prayer lesson for a month. Prayer listening will not be performed to the control group. At the end of one month, the severity of dyspnea, anxiety and spiritual well-being levels of people in both groups will be re-evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 90 individuals (45 experiments, 45 controls) who can be contacted, who have agreed to participate in the study
* who are literate, can speak Turkish
* who have not participated in a similar application of this study before
* who have agreed to participate in the study after being informed about the research
* are 18 years old and over, with a COPD diagnosis will be taken

Exclusion Criteria:

* Individuals with mental and hearing problems, who have lost a family member and someone close to them in the last year
* who are using tranquilizers/antidepressants
* who have experienced a traumatic situation such as divorce will be excluded from the sample.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-05-04 (Actual)

PRIMARY OUTCOMES:
dyspnea 12 scale | 1 month
  as a result of 1-month prayer listening, the severity of dyspnea of the participants in the experimental group decreased. A minimum of 0 and a maximum of 36 points are taken from the scale. The increase in scores indicates that the frequency of dyspnea of patients has increased.
Beck anxiety scale | 1 month
  as a result of listening to prayer for 1 month, the anxiety severity of the participants in the experimental group decreased. A minimum of 0 and a maximum of 63 points are taken from the scale. The increase in scores indicates that the frequency of anxiety of patients has increased.
Spiritual Well-Being Scale | 1 month
  as a result of listening to prayer for 1 month, the spiritual well-being levels of the participants in the experimental group increased. A minimum of 0 and a maximum of 48 points are taken from the scale. An increase in scores indicates an increase in the spiritual well-being of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Gülden Kaygusuz Gülden Kaygusuz, Principal Investigator — Tokat Zile Devlet Hatanesi
Locations (1):
- Zile Devlet Hastanesi, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is not intended to share the data of individual participants.